CLINICAL TRIAL: NCT07112885
Title: Effect of Arthroscopic Microfracture Combined With Stromal Vascular Fraction Therapy on Clinical and Radiological Outcomes in Gonarthrosis: A Prospective Randomized Controlled Trial
Brief Title: Comparison of SVF Injection With and Without Microfracture in Moderate Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Mehmet Yağız Yenigün, Resident Doctor, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IU-ORT-MYY-01
Record Dates: First submitted 2025-08-02; First posted 2025-08-08 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Knee Osteoarthritis (Knee OA)
Keywords: microfracture; Stromal Vascular Fraction; Cartilage Repair; WOMAC; WORMS; Regenerative Medicine
MeSH Terms: conditions — Osteoarthritis, Knee; Fractures, Stress

STUDY DESIGN:
Intervention Model Description: Two-group parallel design: Group A received arthroscopic microfracture combined with stromal vascular fraction injection, while Group B received stromal vascular fraction injection alone.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants were blinded to their treatment allocation throughout the study. Although the operating surgeons were aware of the intervention due to the nature of the surgical procedures, outcome assessment was conducted by an independent radiologist who was blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microfracture Plus SVF Group (Experimental): Participants underwent arthroscopic debridement and microfracture, followed by intra-articular injection of autologous stromal vascular fraction (SVF) derived from adipose tissue.
  Interventions: Procedure: Arthroscopic Microfracture Combined with Autologous SVF Injection
- SVF Only Group (Experimental): Participants underwent only arthroscopic debridement. Following this, autologous SVF derived from adipose tissue was injected intra-articularly, without performing microfracture.
  Interventions: Procedure: Arthroscopic Debridement Followed by Autologous SVF Injection

INTERVENTIONS:
Procedure: Arthroscopic Microfracture Combined with Autologous SVF Injection — This procedure involved arthroscopic debridement and microfracture of the knee joint. After microfracture, autologous SVF, isolated from adipose tissue through mechanical digestion and centrifugation, was administered intra-articularly under sterile conditions
  Arms: Microfracture Plus SVF Group
Procedure: Arthroscopic Debridement Followed by Autologous SVF Injection — This procedure included only arthroscopic debridement of the knee joint. After debridement, autologous SVF, isolated in the same manner from adipose tissue, was injected into the joint space intra-articularly without microfracture.
  Arms: SVF Only Group

SUMMARY:
This prospective, randomized controlled clinical trial aims to evaluate the clinical and radiological effects of combining stromal vascular fraction (SVF) therapy with arthroscopic microfracture in patients with knee osteoarthritis. A total of 50 patients with symptomatic gonarthrosis were randomly assigned to either receive arthroscopic debridement and intra-articular SVF injection alone or SVF injection combined with arthroscopic debridement, microfracture. The primary outcome measures include changes in VAS, WOMAC, and Lysholm scores at 3, 6, 12, and 24 months. Radiological assessment was performed using the Whole-Organ Magnetic Resonance Imaging Score (WORMS) system. The study hypothesis is that the combination therapy will result in superior clinical and cartilage regeneration outcomes compared to SVF treatment alone.

DETAILED DESCRIPTION:
This single-center, prospective, randomized controlled clinical study was conducted to compare the efficacy of stromal vascular fraction (SVF) therapy alone versus SVF therapy combined with arthroscopic microfracture in patients diagnosed with knee osteoarthritis (gonarthrosis). A total of 50 patients with symptomatic medial compartment osteoarthritis, classified as Kellgren-Lawrence grade II-III, were enrolled and randomized into two groups:

Group A (n=25): Participants initially underwent arthroscopic debridement and microfracture, followed by intra-articular injection of autologous stromal vascular fraction (SVF)

Group B (n=25): Participants underwent arthroscopic debridement, after which intra-articular injection of autologous stromal vascular fraction (SVF) was administered. Microfracture was not performed in this group.

SVF was isolated from autologous lipoaspirate obtained via mini-liposuction and processed intraoperatively using a closed system. Arthroscopic microfracture was performed with standard technique, targeting cartilage defects in the medial and lateral femoral condyle.

Clinical evaluations were performed preoperatively and at 3, 6, 12, and 24 months post-intervention using:

Visual Analog Scale (VAS) for pain

Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)

Lysholm Knee Scoring Scale

Radiological outcomes were assessed using 3.0 Tesla MRI and scored with the Whole-Organ Magnetic Resonance Imaging Score (WORMS), focusing on cartilage integrity in predefined regions.

The primary endpoint was the improvement in WOMAC score.Cartilage morphology based on WORMS at 12 and 24 months. Secondary endpoints included changes in Lysholm and VAS scores. Inter-group comparisons were analyzed using appropriate statistical methods with a significance threshold of p < 0.05.

The study aims to explore whether the addition of microfracture to SVF therapy yields superior clinical and structural benefits, potentially guiding future treatment protocols for early to moderate knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage II-III osteoarthritis of the knee
* Patients with a mechanical axis deviation not exceeding 15 mm on the anteroposterior orthoroentgenogram x-ray

Exclusion Criteria:

* Patients with deformities on anteroposterior and lateral x-ray examinations
* Patients with a BMI greater than 35 kg/m2
* Patients diagnosed with secondary gonarthrosis (Rheumatoid arthritis, secondary to trauma)
* Patients with a history of intra-articular injections within the last 6 months
* Patients with a history of knee joint surgery

Ages: 49 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-02-02 (Actual); Primary Completion 2025-04-07 (Actual); Study Completion 2025-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yağız M Yenigün, Principal Investigator — Istanbul University Faculty of Medicine, Topkapi, Turgut Ozal Millet Street, 34093 Fatih/Istanbul
Locations (1):
- Istanbul University Faculty of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nguyen PD, Tran TD, Nguyen HT, Vu HT, Le PT, Phan NL, Vu NB, Phan NK, Van Pham P. Comparative Clinical Observation of Arthroscopic Microfracture in the Presence and Absence of a Stromal Vascular Fraction Injection for Osteoarthritis. Stem Cells Transl Med. 2017 Jan;6(1):187-195. doi: 10.5966/sctm.2016-0023. Epub 2016 Aug 29. PMID 28170179
- [Result] Bisicchia S, Bernardi G, Pagnotta SM, Tudisco C. Micro-fragmented stromal-vascular fraction plus microfractures provides better clinical results than microfractures alone in symptomatic focal chondral lesions of the knee. Knee Surg Sports Traumatol Arthrosc. 2020 Jun;28(6):1876-1884. doi: 10.1007/s00167-019-05621-0. Epub 2019 Jul 11. PMID 31297576

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with moderate knee osteoarthritis were recruited from Istanbul University orthopedics outpatient clinics between 2022-2025. A total of 50 patients were screened and randomized.All participants met inclusion criteria and provided informed consent.
Pre-assignment Details: Seven patients were excluded before assignment due to not meeting eligibility criteria (n=4) or declining participation (n=3).
Period: Overall Study
Arm/Group | Microfracture Plus SVF Group | SVF Only Group
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: A total of 50 participants were analyzed at baseline, with 25 assigned to the Microfracture + SVF group and 25 assigned to the SVF-only group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Microfracture Plus SVF Group | SVF Only Group | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age presented as mean ± standard deviation in years.
  Years | 58.8 (5.6) | 58.6 (5.3) | 58.7 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Number of participants by sex (Female, Male), reported as counts.
  Participants
    Female | 17 | 19 | 36
    Male | 8 | 6 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants] — All participants were recruited from Istanbul University, Istanbul, Turkey.
  Participants
    Turkey | 25 | 25 | 50
Baseline WOMAC Score [Mean (Standard Deviation); unit: Score] — Western Ontario and McMaster Universities Osteoarthritis Index (0-96). Higher scores indicate worse symptoms.
  Score | 50.92 (7.49) | 50.04 (7.38) | 50.48 (7.37)
Baseline Lysholm Score [Mean (Standard Deviation); unit: Score] — Lysholm Knee Scoring Scale (0-100). Higher scores indicate better knee function, with 100 representing normal function and lower scores indicating more severe symptoms.
  Score | 47.20 (5.02) | 47.80 (5.02) | 47.50 (4.97)
Baseline VAS (Pain) [Mean (Standard Deviation); unit: Score] — Visual Analog Scale (VAS) for pain intensity (0-10). Higher scores indicate greater pain.
  Score | 6.56 (1.00) | 6.44 (1.00) | 6.50 (0.99)
Baseline WORMS(Whole-Organ Magnetic Resonance Imaging Score) [Mean (Standard Deviation); unit: Scores on a scale] — The Whole-Organ Magnetic Resonance Imaging Score (WORMS) is a semi-quantitative scoring system used to assess structural integrity of the knee joint in osteoarthritis.
  In this study, only the cartilage subscore was evaluated. Cartilage lesions were graded in 14 anatomical regions of the knee on a scale from 0 to 6 (0 = normal cartilage; 6 = diffuse full-thickness loss). The maximum possible cartilage WORMS subscore is 84, with higher scores indicating more severe cartilage damage.
  Scores on a scale | 68.72 (2.48) | 69.04 (2.62) | 68.88 (2.53)

OUTCOME MEASURES:

1. Primary Outcome: Change in WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index)
Description: The WOMAC index (range: 0-96) is a validated questionnaire evaluating pain, stiffness, and physical function in osteoarthritis patients. Higher scores indicate worse symptoms. This outcome measures change in WOMAC score following SVF therapy with or without microfracture.
Time Frame: Baseline, 3 months, 6 months, 12 months, and 24 months after the intervention
Population: All randomized participants (n=50; 25 in the Microfracture plus SVF group and 25 in the SVF only group) completed the 24-month follow-up and were included in the final analysis. Therefore, the analysis population matches the assigned population.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Microfracture Plus SVF Group | SVF Only Group
Number analyzed (Participants) | 25 | 25
Score
  Outcomes at 3 Months | 49.52 (7.58) | 50.60 (8.64)
  Outcomes at 6 Months | 34.16 (16.32) | 49.96 (7.87)
  Outcomes at 12 Months | 33.88 (5.98) | 47.16 (7.02)
  Outcomes at 24 Months | 33.48 (6.40) | 47.08 (7.68)

2. Primary Outcome: Change in WORMS (Whole-Organ Magnetic Resonance Imaging Score)
Description: The WORMS cartilage subscore (range: 0-84) is a semiquantitative MRI-based system assessing the morphology and integrity of articular cartilage in the knee joint. Higher scores indicate more severe cartilage damage. This outcome specifically evaluates radiological changes in cartilage structure after SVF therapy with or without microfracture.
Time Frame: Baseline and 12,24 months after the intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Microfracture Plus SVF Group | SVF Only Group
Number analyzed (Participants) | 25 | 25
Scores on scale
  Outcomes at 12 Months | 41.28 (2.48) | 68.76 (2.80)
  Outcomes at 24 Months | 40.64 (2.72) | 66.80 (6.25)

3. Secondary Outcome: Change in Lysholm Knee Score
Description: The Lysholm Knee Score (range: 0-100) is a validated tool assessing knee function, including pain, instability, and swelling. Higher scores indicate better knee function.
Time Frame: Baseline, 3 months, 6 months, 12 months, and 24 months after the intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Microfracture Plus SVF Group | SVF Only Group
Number analyzed (Participants) | 25 | 25
Score
  Outcomes at 3 Months | 46.80 (4.76) | 47.6 (5.02)
  Outcomes at 6 Months | 47.40 (5.02) | 46.40 (4.68)
  Outcomes at 12 Months | 82.20 (5.02) | 82.20 (5.02)
  Outcomes at 24 Months | 82.00 (4.08) | 82.40 (5.61)

4. Secondary Outcome: Change in VAS (Visual Analog Scale) for Pain
Description: The VAS for pain (range: 0-10) is a subjective scale assessing pain intensity, where 0 = no pain and 10 = worst imaginable pain. Higher scores indicate worse pain.
Time Frame: Baseline, 3 months, 6 months, 12 months, and 24 months after the intervention
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Microfracture Plus SVF Group | SVF Only Group
Number analyzed (Participants) | 25 | 25
Score
  Outcomes at 3 Months | 5.60 (1.04) | 6.28 (1.06)
  Outcomes at 6 Months | 5.96 (1.17) | 6.16 (1.07)
  Outcomes at 12 Months | 2.76 (0.78) | 5.76 (1.13)
  Outcomes at 24 Months | 2.76 (0.66) | 5.40 (0.91)

ADVERSE EVENTS:
Time Frame: From the time of intervention until 24 months follow-up.
Description: Adverse events were systematically monitored throughout the 24-month follow-up using scheduled clinic visits and patient-reported outcome assessments.
Arm/Group | Microfracture Plus SVF Group | SVF Only Group
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

LIMITATIONS AND CAVEATS:
The study is limited by its 24-month follow-up, without long-term data. Cartilage quality was assessed indirectly with WORMS scores, and variability in SVF composition across patients may have influenced outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2025-09-19): https://cdn.clinicaltrials.gov/large-docs/85/NCT07112885/Prot_000.pdf
  • Informed Consent Form (2025-09-12): https://cdn.clinicaltrials.gov/large-docs/85/NCT07112885/ICF_001.pdf